CLINICAL TRIAL: NCT06763458
Title: Balloon Angioplasty for Minor Unstable Stroke With IntraCranial Atherosclerosis Stenosis (BAMUS-ICAS): a Prospective, Randomized, Multi-center Study
Brief Title: Balloon Angioplasty for Minor Unstable Stroke With IntraCranial Atherosclerosis Stenosis (BAMUS-ICAS)
Acronym: BAMUS-ICAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y(2024)262
Record Dates: First submitted 2024-12-22; First posted 2025-01-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: stroke; Submaximal balloon angioplasty; early neurological deterioration; Intracranial atherosclerotic stenosis
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBA group (Experimental): Receiving SBA plus best medical therapy
  Interventions: Procedure: Submaximal balloon angioplasty
- Control group (No Intervention): Receiving best medical therapy

INTERVENTIONS:
Procedure: Submaximal balloon angioplasty — The goal of submaximal balloon angioplasty is to use the balloon to improve the stenosis of the criminal artery by more than 20%.
  Arms: SBA group

SUMMARY:
Intracranial atherosclerotic stenosis (ICAS) is a common cause of stroke, especially in East and South Asia, and is significantly associated with stroke recurrence and early neurological deterioration (END) despite aggressive medical management. Minor stroke (National Institutes of Health Stroke, NIHSS score ≤ 5) patients with ICAS often has higher risk of END. The early realization of blood flow patency is closely related to the improvement of patient outcomes. Submaximal balloon angioplasty (SBA) as a safer and simpler intervention which can improve cerebral blood flow. Thus, SBA may be an effective strategy for preventing END in acute ischemic stroke patients with ICAS.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age;
2. Minor ischemic stroke within 1 week of onset (NIHSS≤5);
3. Have received the best drug treatment (dual antibody, anti-plate combined with anticoagulation), but symptoms still have measurable fluctuations or progression (NIHSS increased by at least 1 point);
4. Symptoms fluctuate to the time of receiving balloon dilation within 24 hours;
5. The etiology was considered to be severe stenosis of the responsible vessels due to intracranial arteriosclerosis (70-99% stenosis), or perforator artery disease with severe stenosis of the carrier artery (confirmed by MRA, CTA or DSA);
6. Patients with first onset or past onset without sequelae such as limb paralysis should not affect the score of this NIHSS, and mRS Score of patients with past onset should be less than 2 points;
7. Patients or family members sign informed consent.

Exclusion Criteria:

1. Patients who have developed large intracranial vessel occlusion;
2. Intracranial hemorrhagic diseases in the past 3 months: cerebral hemorrhage, subarachnoid hemorrhage, etc.;
3. Non-atherosclerotic disease-related stenosis: arterial dissection, moya-moya disease, arterioinflammatory disease, etc.
4. Clotting disorders or systemic bleeding tendency or platelets less than 100,000;
5. Complicated with serious infection or liver, kidney and other serious diseases;
6. Patients with severe inability to control hypertension (systolic blood pressure >200mmHg or diastolic blood pressure >110mmHg);
7. Women who are pregnant, have a pregnancy plan or are breastfeeding;
8. Complicated with other serious diseases, life expectancy < 6 months; Other conditions deemed inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of early neurological deterioration (NIHSS score increase of 4 points or more) | at 24±8 hours

SECONDARY OUTCOMES:
The decrease of NIHSS score | at 24±8 hours
The decrease of NIHSS score | at 10±2 days
Proportion of early neurological improvement (NIHSS score decline of 4 points or 0) | at 24±8 hours
Proportion of patients with modified Rankin Score 0 to 1 | at 90±7 days
Proportion of patients with modified Rankin Score 0 to 2 | at 90±7 days
Distribution of patients with modified Rankin Score | at 90±7 days
the occurence of stroke or other cardiovascular events | at 90±7 days
ischemic stroke in the culprit artery territory | at 90±7 days
Incidence of symptomatic intracranial hemorrhage (ECASS-III criteria) | at 24±8 hours
Proportion of occurrence of cerebral parenchymal hemorrhage types (PH1) and (PH2) | at 24±8 hours
Proportion of serious adverse events | at 24±8 hours
Proportion of all-cause deaths | at 10±2 days
Complications associated with endovascular therapy | at 24±8 hours, at 10±2 days, at 90±7 days

OTHER OUTCOMES:
Changes in cortical oxygen saturation | at 24±8 hours
Changes of cerebral blood flow autoregulation function | at 24±8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: No